CLINICAL TRIAL: NCT05370664
Title: Performance of Novel Bed Side Scores as Predictors of Hospital Outcome in Acute Exacerbation of Chronic Obstructive Pulmonary Disease Among Women; Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Essmat Hussien, Assistant Lecturer of chest diseases and tuberculosis, Assiut University
Other Study IDs: Mortality outcome in COPD
Record Dates: First submitted 2022-05-07; First posted 2022-05-11 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: COPD Exacerbation
Keywords: NIVO, DECAF, HACOR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female COPD
- Male COPD

SUMMARY:
* Assess predictors of mortality in COPD exacerbation between men and women.
* Evaluate the clinical outcomes in acute exacerbation of COPD in women.
* Evaluate the validity of new scoring systems ( NIVO, DECAF, HACOR ) as a predictor for hospital outcome in acute exacerbation of COPD.
* Compare these new scoring system with the most widely used APACHE IV.
* Assessment of serum level of granulocyte colony stimulating factor ( GM-CSF) in detecting the severity of COPD exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AECOPD leading to hypoxemia, hypercapnia and respiratory acidosis with pH < 7.35 and PaCO2 > 45 mm of Hg will be admitted to the respiratory intensive care unit (ICU) for NIV or the ward will be eligible for inclusion and not in need for mechanical ventilation

Exclusion Criteria:

* Requirement for emergency intubation.
* Other contraindications to NIPPV including cardiac or respiratory arrest; nonrespiratory organ failure (eg, severe encephalopathy, severe gastrointestinal bleeding, hemodynamic instability with or without unstable cardiac angina); facial surgery or trauma; upper-airway obstruction; inability to protect the airway and/or high risk of aspiration; and inability to clear secretions.(6)
* Age < 35 years.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients enrolled in the study will be subjected to the following:
  A- Careful History Taking and clinical examination.
  B- Laboratory investigations which include :
  I. Complete blood count. II. Arterial blood gas. III. Liver & kidney function tests. IV. Blood sugar level & serum electrolytes. V. Serum granulocyte colony-stimulating factor ( GM-CSF)
  C- Severity of illness assessed by:
  I. NIVO Score ( Non-invasive outcomes score )
  II. DECAF Score
  III. HACOR Score
  IV. ( Acute physiology and chronic health evaluation ) APACHE IV Score. 200 patients (100 females, 100 males) with acute exacerbation of COPD will be admitted to the RICU will be observed as regards temperature, blood pressure, respiratory rate, pulse, oxygen saturation, and arterial blood gas will be obtained on NIV.
  colony-stimulating factor will also be assessed on the first day of admission and after weaning from NIV.
Sampling Method: Probability Sample
Enrollment: 203 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Mortality rate among COPD patients hospitalized due to acute exacerbation. | 28 days from admissiom
  Assessment of mortality with different scoring systems in acute exacerbation of COPD
Early prediction of NIV failure. | 48 hours from ICU admission
  Using NIVO score for Acute exacerbaion of COPD Non-invasive ventilation outcomes score is considered to be Low risk ( 0-2) Moderate risk (3-4) High risk (5-6) Very high risk ( 7-9)
Assessment of GM-CSF as a biomarker for successful therapy in acute exacerbation of COPD. | baseline
  Assessment of granulocyte colony stimulating factor by ELISA test in acute exacerbation of COPD

SECONDARY OUTCOMES:
Assisted ventilation days. | Baseline
  Estimating the number of days required for either non-invasive or invasive mechanical ventilation

REFERENCES:
- [Background] Halpin DMG, Criner GJ, Papi A, Singh D, Anzueto A, Martinez FJ, Agusti AA, Vogelmeier CF. Global Initiative for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease. The 2020 GOLD Science Committee Report on COVID-19 and Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2021 Jan 1;203(1):24-36. doi: 10.1164/rccm.202009-3533SO. PMID 33146552
- [Background] Chakrabarti A, Mar JS, Choy DF, Cao Y, Rathore N, Yang X, Tew GW, Li O, Woodruff PG, Brightling CE, Grimbaldeston M, Christenson SA, Bafadhel M, Rosenberger CM. High serum granulocyte-colony stimulating factor characterises neutrophilic COPD exacerbations associated with dysbiosis. ERJ Open Res. 2021 Aug 2;7(3):00836-2020. doi: 10.1183/23120541.00836-2020. eCollection 2021 Jul. PMID 34350278
- [Background] Jenkins CR, Chapman KR, Donohue JF, Roche N, Tsiligianni I, Han MK. Improving the Management of COPD in Women. Chest. 2017 Mar;151(3):686-696. doi: 10.1016/j.chest.2016.10.031. Epub 2016 Nov 2. PMID 27816445
- [Background] Duan J, Wang S, Liu P, Han X, Tian Y, Gao F, Zhou J, Mou J, Qin Q, Yu J, Bai L, Zhou L, Zhang R. Early prediction of noninvasive ventilation failure in COPD patients: derivation, internal validation, and external validation of a simple risk score. Ann Intensive Care. 2019 Sep 30;9(1):108. doi: 10.1186/s13613-019-0585-9. PMID 31565779
- [Background] Hartley T, Lane ND, Steer J, Elliott MW, Sovani MP, Curtis HJ, Fuller ER, Murphy PB, Shrikrishna D, Lewis KE, Ward NR, Turnbull CD, Hart N, Bourke SC. The Noninvasive Ventilation Outcomes (NIVO) score: prediction of in-hospital mortality in exacerbations of COPD requiring assisted ventilation. Eur Respir J. 2021 Aug 12;58(2):2004042. doi: 10.1183/13993003.04042-2020. Print 2021 Aug. PMID 33479109
- [Background] Steer J, Gibson J, Bourke SC. The DECAF Score: predicting hospital mortality in exacerbations of chronic obstructive pulmonary disease. Thorax. 2012 Nov;67(11):970-6. doi: 10.1136/thoraxjnl-2012-202103. Epub 2012 Aug 15. PMID 22895999